CLINICAL TRIAL: NCT05061290
Title: The Potential of Food to Food Fortification to Improve Iron Bioavailability From Cereal-based Foods
Brief Title: Iron Bioavailability From Cereal-based Foods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Purdue University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bruce R. Hamaker, Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-2019-764
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Iron Bioavailability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control Porridge (Experimental): Wholegrain maize flour, Mango powder, Carrot powder, Ferrous sulfate, Corn starch
  Interventions: Other: Control Porridge
- Reference Porride A (Experimental): Wholegrain maize flour, Mango powder, Carrot powder, Ferrous sulfate, Ascorbic acid, Corn starch
  Interventions: Other: Reference Porridge A
- Test Porridge B (Experimental): Wholegrain maize flour, Moringa leaf powder, Mango powder, Carrot powder, Corn starch
  Interventions: Other: Test Porridge B
- Test Porridge C (Experimental): Wholegrain maize flour, Baobab fruit powder, Mango powder, Carrot powder, Ferrous sulfate, Corn starch
  Interventions: Other: Test Porridge C
- Test Porridge D (Experimental): Wholegrain maize flour, Baobab fruit powder, Moringa leaf powder, Mango powder, Carrot powder
  Interventions: Other: Test Porridge D

INTERVENTIONS:
Other: Control Porridge — Maize porridge containing 54Fe as iron sulfate
  Arms: Control Porridge
Other: Reference Porridge A — Maize porridge counting 58Fe as iron sulfate with ascorbic acid
  Arms: Reference Porride A
Other: Test Porridge B — Maize porridge containing 57Fe and fortified with Moringa leaf powder as iron source
  Arms: Test Porridge B
Other: Test Porridge C — Maize porridge containing 57Fe and fortified with Boabab fruit powder as iron source
  Arms: Test Porridge C
Other: Test Porridge D — Maize porridge containing 54Fe and fortified with Moringa leaf and Baobab fruit powder as iron source
  Arms: Test Porridge D

SUMMARY:
Iron-deficient anemia is a chronic problem in sub-Saharan Africa and other developing areas of the world. From our previous research, the investigators have shown that certain local plant foods in Kenya and Senegal have an unusual action of improving in vitro iron bioaccessibility (nearly doubling the low value obtained in cereals). The investigators will assess absorption of stable isotopes of iron (57Fe, 54Fe and 58Fe) extrinsically labeled in a serving of porridge fortified with various combinations of moringa, baobab, mango, carrot and standard fortificant iron sulfate and the enhancer ascorbic acid.

DETAILED DESCRIPTION:
To better understand the potential for leveraging traditional plant-based ingredients in local fortification efforts in Africa, the proposed study will focus on assessment of acute iron bioavailability in participants consuming instant blended cereal porridges produced using whole grain white maize, with provitamin A (e.g. carrots/mango), moringa leaf powder and baobab fruit powder in specific combinations. The investigators hypothesize that: food-to-food fortified cereal-based porridge with with African baobab fruit and moringa leaf powder will effectively improve iron density and bioavailability in human participants as compared to a "gold standard" fortification (iron sulphate and ascorbic acid).

A randomized crossover design with 4 different white maize cereal-based porridges and a reference control porridge (with matching macronutrient contents) will be used, allowing each participant to serve as their own control. Porridges are designed to specifically compare: (1) Food to food fortification versus standard fortifications and (2) the ability of baobab fruit pulp to enhance iron absorption from both natural and standard sources. The porridges will be composed of locally sourced ingredients including: whole grain white maize, a pro-vitamin A source (oil and available vegetables e.g. carrot and mango) baobab fruit powder and moringa leaf powder.

The enrolled participants will come into the clinic 6 times to consume porridges or have blood drawn. Four times blood (1 for screening, 3 for study) will be drawn to determine the amount of the different forms of iron in participant's blood. On each day of porridge consumption (each visit except the final visit on Day 33), they will consume 2 x 350 g porridge meals and stay 90 mins after the participant has finished each of the meals, and then leave and come back to repeat for a total of 4 hours. After two weeks they will return to the clinic and the investigators will ask to draw some more blood to see if they have absorbed any of the different forms of iron. They will then have the next porridge. Importantly for each visit for both blood draws and the porridge consumption the participants will have to fast the previous night, so no food or beverages like tea or coffee can be consumed (only water allowed). During 5 visits when they will eat two portions of porridge during the day and will have to stay at the facility for 90 mins after each porridge consumption. During the last visit (Day 33), participants will need to give a blood sample, which will take about half an hour. Blood collected during these visits will be used to measure isotopic iron absorbed from the porridges.

ELIGIBILITY:
Inclusion:

* Female 18-65 Y
* BMI 18.5-25 kg/m2
* Stable weight past 3 month (+/- 2.5kg)
* Clinically normal blood profiles
* Fasting blood glucose < 110 and CRP below 3 mg/L

Exclusion:

* Smokers and vapers
* No heavy alcohol consumption (>2 drinks per day)
* Diabetic
* Presence of metabolic of intestinal disorder including lipid malabsorption or lactose intolerance
* Male sex
* Pregnant
* Lactating
* Long term use of medications
* Blood donation in past 4 months
* Previous participation in iron stable isotope bioavailability study
* Following a weight reduction program or having one in past 3 months
* Peri- or post-menopausal
* Acute or chronic disease
* Hypertension

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Iron absorption | Acute study but blood measurement to occur following 14 daysof acute consumption
  Assessment whole blood for isotopic iron absorption from individual meals

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers